CLINICAL TRIAL: NCT00295529
Title: GenetiKiT: Evaluation of the Impact of a Multifaceted Intervention to Enhance the Delivery of Genetics Services by Family Physicians.
Brief Title: GenetiKiT: Evaluation of an Educational Intervention on the Delivery of Genetics Services by Family Physicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, June Carroll, Associate Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 04-0109-E
Record Dates: First submitted 2006-02-09; First posted 2006-02-23 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Breast Neoplasm
Keywords: Primary health care; Breast neoplasm; Education
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multifaceted Educational Intervention (Experimental): Intervention group received an interactive workshop, portfolio of primary care appropriate genomics tools, and Gene Messengers
  Interventions: Behavioral: Multifaceted educational intervention
- No education (No Intervention): Educational materials at end of study

INTERVENTIONS:
Behavioral: Multifaceted educational intervention — Educational materials available at end of study
  Arms: Multifaceted Educational Intervention

SUMMARY:
There is an urgent need for a knowledge translation strategy to facilitate the integration of genetics into family medicine, to improve the low knowledge base of most Canadian family physicians, ensure that the needs are met of those in the population who could benefit from genetic assessment, and facilitate evidence-based decision-making in the face of increasing patient demand.

We have developed a multi-faceted intervention incorporating three distinct knowledge translation strategies: interactive educational sessions, a portfolio of tools for use in clinical practice and an innovative, efficient, information technology-based knowledge service designed to provide timely ("just-in-time") information which reflects both topical genetics issues and the pattern of users' queries (a so-called "push-pull" approach).

We hypothesize that a multi-faceted knowledge translation intervention will improve the delivery of genetics services by family physicians.

DETAILED DESCRIPTION:
The intervention will be evaluated using a randomized controlled trial, in which family physicians will be allocated to receive the active or control interventions, with pre-intervention data collected 1 month prior, and post-intervention outcome data 6 months following the intervention.

A list of practicing family physicians will be obtained from the chiefs of Family Medicine at local hospitals in Toronto, Ottawa, Timmins, and Thunder Bay. We will develop a sampling frame for each site reflecting the proportion of solo and group practitioners in the community. A statistician independent of the study will generate a random number sequence to allocate practitioners to the control or intervention groups. There is a potential danger of contamination if two family physicians are recruited from the same group practice and randomized to different study arms, therefore only one physician per practice will be invited to participate in the study. Once one family physician has been recruited from a practice, all other physicians from the same practice will be deleted from the sampling frame.

Our intervention has three components: an interactive educational workshop, a portfolio of tools for family physicians to use in their day to day clinical practice, and a new IT-based knowledge service.

The workshop will deal with practical medical genetics knowledge, risks, benefits and limitations of genetic testing including psychosocial risks, confidentiality and insurance issues as well as a critical appraisal framework by which to assess genetic tests. The workshop will be 60 minutes in length and offered at several times and dates to facilitate attendance. The College of Family Physicians of Canada educational credit of 1 hour is available for participation in this project.

Several tools will be presented at the workshop:

A) A family history tool B) Genetics Pearls C) Physician risk triage and management cards for familial cancer covering risk assessment and management of hereditary breast and colorectal cancer.

D) A table outlining the possible consequences of genetic test results E) Patient information aids to help patients self-identify their risk of hereditary cancer F) GeneMessenger is designed primarily to address knowledge gaps about specific genetics issues in the news, about which family physicians may feel ill-equipped to form confident opinions. The research team will scan the mainstream print media for headlines or stories that relate to medical genetics discoveries or topics. Supported by a geneticist and an expert family physician, a genetic counselor will appraise the discoveries, tests or interventions for their relevance to family practice. She will prepare a definitive short review for participants within 1-2 weeks, but, where appropriate and possible, will prepare a preliminary comment for rapid communication within 1-2 days. Communication will be by email or fax as chosen by the participant. Family physicians will be able to contact the service to suggest questions or topics they would like to see addressed. This service will not provide professional advice on specific cases or patients and referrals to genetics clinics would continue in the usual fashion. Physicians would be free to seek telephone advice from geneticists or counselors regarding specific patients but these would not be addressed as part of this service.

Data will be collected one month before and six months after the intervention by postal survey to the participating physicians. Changes in intention to refer to genetics services in response to 10 clinical vignettes will be compared between the control and intervention group.

ELIGIBILITY:
Inclusion Criteria:

* family physicians in active practice
* practicing in one of the study communities

Exclusion Criteria:

* only one family physician per group practice
* physicians participating in one of the investigator's ongoing primary care genetics projects

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2005-04; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Intention to refer to genetic services based on clinical vignettes | 1 year

SECONDARY OUTCOMES:
Self-efficacy | 1 year
Recall and understanding of information | 1 year
Perceived decisional conflict | 1 year
Physicians' perceptions of the value of the components of the intervention | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: June C Carroll, MD, Principal Investigator — Mount Sinai Hospital University of Toronto; Judith E Allanson, MD FRCP, Principal Investigator — Children's Hospital of Eastern Ontario; Brenda J Wilson, BSc MSc MB, Principal Investigator — University of Ottawa
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Carroll JC, Wilson BJ, Allanson J, Grimshaw J, Blaine SM, Meschino WS, Permaul JA, Graham ID. GenetiKit: a randomized controlled trial to enhance delivery of genetics services by family physicians. Fam Pract. 2011 Dec;28(6):615-23. doi: 10.1093/fampra/cmr040. Epub 2011 Jul 10. PMID 21746696